CLINICAL TRIAL: NCT04801615
Title: Demographic Characteristics, Symptoms, Treatment and Mortality of Patients With Necrotizing Soft Tissue Infections
Brief Title: Characteristics of Patients With Necrotizing Soft Tissue Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Per Gundtoft, Principal Investigator, Consultant, PhD, Aarhus University Hospital
Other Study IDs: ICD_20201212
Record Dates: First submitted 2020-12-23; First posted 2021-03-17 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Necrotizing Soft Tissue Infection
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surgery — All patients in the database undergo surgery due to a suspicion of necrotizing soft tissue infections

SUMMARY:
To study the demographic characteristic of patients with necrotizing soft tissue infections.

DETAILED DESCRIPTION:
At Aarhus University Hospital, Denmark, all patients with necrotizing soft tissue infections will be registered in a database in order to be able to describe their symptoms, demographic variables and thier treatment (surgery, time to surgery, antibiotics, intensive care unit, laboratory data etc).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with necrotizing soft tissue infections and treated at Aarhus Universital Hospital

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to Aarhus University Hospital with necrotizing soft tissue infections, either diagnosed prior to arriving to the hospital or diagnosed in the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients that dies within 1 year following admission date | 12 months following admission date
  The risk of death within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: per gundtoft, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
We do not plan to share this with other researchers.